CLINICAL TRIAL: NCT00257192
Title: Six Week, Double-Blind, Placebo Controlled Phase III Trial Evaluating The Efficacy, Safety And Pharmacokinetics Of Flexible Doses Of Oral Ziprasidone In Adolescent Subjects With Schizophrenia
Brief Title: Safety And Efficacy Of Ziprasidone In Adolescents With Schizophrenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Please see Detailed Description for termination reason.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A1281134
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Results first posted 2010-04-13 (Estimated); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Schizophrenia
Keywords: Adolescent Subjects With Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — ziprasidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2.0 (Placebo Comparator)
  Interventions: Drug: placebo
- 1.0 (Active Comparator)
  Interventions: Drug: Ziprasidone oral capsules

INTERVENTIONS:
Drug: placebo — Placebo matching the oral ziprasidone capsules of 20 mg, 40 mg, 60 mg, and 80 mg strength or matching placebo. Subjects will be dosed daily for 6 weeks using a flexible dose design with a minimal dose range of 40mg twice a day (BID) to a maximum dose range of 80 mg BID. For subjects weighing <45 kg, the doses will range from 20 mg BID to 40 mg BID.
  Arms: 2.0
Drug: Ziprasidone oral capsules — Oral ziprasidone capsules of 20 mg, 40 mg, 60 mg, and 80 mg strength or matching placebo. Subjects will be dosed daily for 6 weeks using a flexible dose design with a minimal dose range of 40mg BID to a maximum dose range of 80 mg BID. For subjects weighing <45 kg, the doses will range from 20 mg BID to 40 mg BID.
  Other Names: Geodon, Zeldox
  Arms: 1.0

SUMMARY:
The purpose of this study is to determine if flexibly-dosed ziprasidone is safe and effective for the treatment of adolescents (ages 13-17) with schizophrenia

DETAILED DESCRIPTION:
Termination Reason: On March 24, 2009, Pfizer Inc. stopped late stage Geodon pediatric clinical trials in schizophrenia (A1281134 - placebo controlled; A1281135 - open label). As recommended by the DSMB, these studies were stopped due to lack of efficacy. No safety concerns were identified.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria for schizophrenia: Current symptoms were to be present for at least 7 days before screening.
* At the Screening and Baseline visits, subjects must have had a Brief Psychiatric Rating Scale - Anchored score ≥35 and a score of ≥4 on at least 1 of the following items: unusual thought content (i.e., delusions), hallucinations, suspiciousness, or conceptual disorganization.
* Age 13 - 17 years

Exclusion Criteria:

* Imminent risk of suicide or homicide, as judged by the site investigator
* Any history of serious or unstable medical illness, including risk for QT prolongation

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 284 (Actual)
Dates: Start 2006-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (72):
- United States (37):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Stanford, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Altamonte Springs, Florida
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, North Miami, Florida
  - Pfizer Investigational Site, Orange City, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Tavares, Florida
  - Pfizer Investigational Site, Smyrna, Georgia
  - Pfizer Investigational Site, Tucker, Georgia
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Des Plaines, Illinois
  - Pfizer Investigational Site, Oakbrook Terrace, Illinois
  - Pfizer Investigational Site, Schaumburg, Illinois
  - Pfizer Investigational Site, Pikesville, Maryland
  - Pfizer Investigational Site, Towson, Maryland
  - Pfizer Investigational Site, Clinton Township, Michigan
  - Pfizer Investigational Site, Meridian, Mississippi
  - Pfizer Investigational Site, Bridgeton, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Arlington, Texas
  - Pfizer Investigational Site, DeSoto, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, Bothell, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
  - Pfizer Investigational Site, West Allis, Wisconsin
- Colombia (2):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Bogota, Cundinamarca
- Pfizer Investigational Site, San José, Costa Rica
- India (9):
  - Pfizer Investigational Site, Vijaywada, Andhra Pradesh
  - Pfizer Investigational Site, Visakhapatnam, Andra Pradesh/India
  - Pfizer Investigational Site, Ahmedabad, Guj
  - Pfizer Investigational Site, Mangalore, Karnataka
  - Pfizer Investigational Site, Aurangabad, Maharashtra
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, Ludhiana, Punjab
  - Pfizer Investigational Site, Chennai, Tamil Nadu
- Malaysia (2):
  - Pfizer Investigational Site, Kubang Kerian, Kelantan
  - Pfizer Investigational Site, Kuala Lumpur
- Pfizer Investigational Site, Lima, Peru
- Russia (9):
  - Pfizer Investigational Site, Kazan'
  - Pfizer Investigational Site, Khotkovo, Moscow Region
  - Pfizer Investigational Site, Lipetsk Region
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Nizhny Novgorod
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Saratov
  - Pfizer Investigational Site, Tver'
  - Pfizer Investigational Site, Yaroslavl
- Pfizer Investigational Site, Singapore, Singapore
- Ukraine (10):
  - Pfizer Investigational Site, Simferopol, Autonomous Republic of Crimea
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Donetsk
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Luhansk
  - Pfizer Investigational Site, Lviv
  - Pfizer Investigational Site, Odesa
  - Pfizer Investigational Site, Poltava
  - Pfizer Investigational Site, Vinnytsia

REFERENCES:
- [Derived] Findling RL, Cavus I, Pappadopulos E, Vanderburg DG, Schwartz JH, Gundapaneni BK, DelBello MP. Ziprasidone in adolescents with schizophrenia: results from a placebo-controlled efficacy and long-term open-extension study. J Child Adolesc Psychopharmacol. 2013 Oct;23(8):531-44. doi: 10.1089/cap.2012.0068. Epub 2013 Oct 10. PMID 24111983
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281134&StudyName=Safety%20and%20efficacy%20of%20ziprasidone%20in%20adolescents%20with%20schizophrenia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A planned interim analysis resulted in recommendation from Data Safety Monitoring Board (DSMB) to terminate study due to futility per the interim analysis charter (p-value = 0.9840). Only one active subject in the study was affected by this decision.
Pre-assignment Details: Screening visit followed by a 1 to 10 day period to allow for wash-out of exclusionary medications.
Groups:
- Ziprasidone: Oral (PO) capsules administered twice daily (BID) with meals; titrated from a starting dose of 20 milligrams per day (mg/day) over 2 weeks with dose increases of 20 mg/day every second day up to a target dose range of 120 to 160 mg/day for subjects with body weight ≥ 45 kilograms (kg); target dose for subjects with body weight < 45 kg is 60 to 80 mg/day. After titration dose is attained, flexible dosing range of 80 to 160 (if body weight ≥ 45 kg) or 40 to 80 mg/day (if body weight < 45 kg) for duration of the study.
- Placebo: Placebo matching ziprasidone administration: PO capsules administered BID) with meals; titrated from a starting dose of 20 mg/day over 2 weeks with dose increases of 20 mg/day every second day up to a target dose range of 120 to 160 mg/day for subjects with body weight ≥ 45 kg; target dose for subjects with body weight < 45 kg is 60 to 80 mg/day. After titration dose is attained, flexible dosing range of 80 to 160 (if body weight ≥ 45 kg) or 40 to 80 mg/day (if body weight < 45 kg) for duration of the study.
Period: Overall Study
Arm/Group | Ziprasidone | Placebo
Started | 193 | 91 (Includes 1 subject randomized but not treated)
Received Study Treatment | 193 | 90
Completed | 135 | 52
Not Completed | 58 | 39
Not completed — Adverse Event | 21 | 10
Not completed — Laboratory abnormality | 1 | 1
Not completed — Lost to Follow-up | 3 | 3
Not completed — Insufficient clinical response | 18 | 18
Not completed — Withdrawal by Subject | 14 | 2
Not completed — Randomized but not treated | 0 | 1
Not completed — Study terminated by sponsor | 1 | 0
Not completed — Miscellaneous | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ziprasidone | Placebo | Total
Number analyzed (Participants) | 193 | 90 | 283
Age, Customized [Number; unit: participants]
  >12 years and <13 years at start of treatment | 4 | 0 | 4
  Between 13 and 17 years | 189 | 90 | 279
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.3 (1.4) | 15.4 (1.4) | 15.3 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 28 | 112
  Male | 109 | 62 | 171
Ethnicity [Number; unit: participants]
  Hispanic / Latino | 21 | 9 | 30
  Not Hispanic / Latino | 172 | 81 | 253
Race [Number; unit: particpants]
  White | 116 | 60 | 176
  Black | 17 | 2 | 19
  Asian | 38 | 17 | 55
  Hispanic | 9 | 3 | 12
  Other | 13 | 8 | 21
Tanner adolescent pubertal self-assessment: Breast (females) [Number; unit: particpants] — At baseline, subjects self-administer a gender appropriate Tanner Adolescent Pubertal Staging Questionnaire to document the stage of development of secondary sexual characteristics. Female pubertal development staged by pubic hair development and breast size; males pubertal development staged by size of the genitalia and development of pubic hair. Rated in 5 stages: stage 1 (no development) to 5 (adult-like development in quantity and size).
  particpants
    Stage 1 | 0 | 1 | 1
    Stage 2 | 6 | 3 | 9
    Stage 3 | 16 | 4 | 20
    Stage 4 | 35 | 11 | 46
    Stage 5 | 25 | 9 | 34
    Not applicable | 109 | 62 | 171
    Missing (not answered) | 2 | 0 | 2
Tanner adolescent pubertal self-assessment: Genitalia (males) [Number; unit: participants] — At baseline, subjects self-administer a gender appropriate Tanner Adolescent Pubertal Staging Questionnaire to document the stage of development of secondary sexual characteristics. Female pubertal development staged by pubic hair development and breast size; males pubertal development staged by size of the genitalia and development of pubic hair. Rated in 5 stages: stage 1 (no development) to 5 (adult-like development in quantity and size).
  participants
    Stage 1 | 0 | 1 | 1
    Stage 2 | 9 | 3 | 12
    Stage 3 | 25 | 16 | 41
    Stage 4 | 57 | 26 | 83
    Stage 5 | 18 | 16 | 34
    Not applicable | 82 | 28 | 110
    Missing (not answered) | 2 | 0 | 2
Tanner adolescent pubertal self-assessment: Pubic hair (females and males) [Number; unit: participants] — At baseline, subjects self-administer a gender appropriate Tanner Adolescent Pubertal Staging Questionnaire to document the stage of development of secondary sexual characteristics. Female pubertal development staged by pubic hair development and breast size; males pubertal development staged by size of the genitalia and development of pubic hair. Rated in 5 stages: stage 1 (no development) to 5 (adult-like development in quantity and size).
  participants
    Stage 1 | 0 | 3 | 3
    Stage 2 | 13 | 7 | 20
    Stage 3 | 36 | 13 | 49
    Stage 4 | 90 | 43 | 133
    Stage 5 | 52 | 24 | 76
    Missing (not answered) | 2 | 0 | 2
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 164.9 (10.1) | 167.8 (10.0) | 165.8 (10.1)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 61.2 (15.5) | 64.3 (15.7) | 62.2 (15.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Brief Psychiatric Rating Scale - Anchored (BPRS-A) Total Score at Week 6
Description: BPRS-A: 18-item clinician rated scale to assess somatic concern, anxiety, emotional withdrawal, disorganization, hallucinatory behavior, guilt feelings, suspiciousness, disorientation, tension, mannerisms, posturing, grandiosity, depressive mood, hostility, motor retardation, uncooperativeness, unusual thought content, blunted affect, and excitement. Ratings anchored to improve consistency for a single rater over time or between raters. Items rated on 7-point scale 0 (not present) to 6 (extremely severe). Total score=sum of items (range 0 to 108); higher scores indicate increased pathology.
Time Frame: Baseline, Week 6
Population: Intent to treat (ITT): all randomized subjects who had baseline measurements, took at least 1 dose of study medication, and had at least 1 post-baseline visit. N=number of subjects with analyzable data at post-baseline observation.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 189 | 87
scores on a scale | -14.16 (0.78) | -12.35 (1.05)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Sample size for 85% power 2-tailed 0.05 significance level based on expected difference of -5 with average within-group standard deviation=13 was 276 subjects (2 to 1 ratio of enrollment: 184 ziprasidone, 92 placebo). Interim analysis at 60 percent (%) enrollment (ITT population): may stop trial early for efficacy (2-sided p-value less than (<) 0.0124) or for futility (2-sided p-value greater than (>) 0.4772; The final analysis is to employ a 2-sided p-value <0.0462; Test type: Superiority or Other; p = 0.1530, ANCOVA — Mixed effects repeated measures (MMRM) analysis of covariance model with subject as random effect, treatment, region, visit and visit-by-treatment interaction as fixed effects and baseline score as a covariate; P-value for final analysis is to be adjusted due to planned interim analysis (0.0462); Least squares mean = -1.80, 95% CI 2-sided [-4.28 to 0.67], Standard Error of Mean 1.26

2. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S) Score at Week 6
Description: CGI-S: single-item clinician rated scale to rate the severity of a subject's illness over time. Scores range from 1 (normal, not at all ill) to 7 (among the most severely ill subjects); higher score indicates more affected.
Time Frame: Baseline, Week 6
Population: ITT; N=number of subjects with analyzable data at post-baseline observation.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 190 | 87
scores on a scale | -1.05 (0.08) | -0.84 (0.12)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Difference from placebo; Test type: Superiority or Other; p = 0.1289, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Hochberg procedure was applied to p-value to preserve type I error in the analysis of key secondary endpoints (PANSS total score and CGI-S); Least squares mean = -0.21, 95% CI 2-sided [-0.48 to 0.06], Standard Error of Mean 0.14

3. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) - Total Score at Week 6
Description: PANSS: 30-item clinician-rated scale to measure severity of psychopathology (16 items); positive scale (7 items); negative scale (7 items); summarized as positive score, negative score, and total score. Items scored on anchored Likert scale rated 1 (absent symptoms) to 7 (extreme); scores above 1 indicate clinical symptom is present; scores from 2 to 7 indicate increased severity. Total score range 30 to 210: higher score indicates greater severity.
Time Frame: Baseline, Week 6
Population: ITT; N=number of subjects with analyzable data at post-baseline observation.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 183 | 86
scores on a scale | -23.58 (1.42) | -21.01 (1.73)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Total score: difference from placebo; Test type: Superiority or Other; p = 0.1987, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 2, analysis 1]; Least squares mean = -2.57, 95% CI [-6.50 to 1.36], Standard Error of Mean 2.00

4. Secondary Outcome: Change From Baseline in PANSS: Positive and Negative Subscales at Week 6
Description: as for outcome 3
Time Frame: Baseline, Week 6
Population: ITT; N=number of subjects with analyzable data at post-baseline observation.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 183 | 86
scores on a scale
  Positive score | -7.22 (0.44) | -5.88 (0.56)
  Negative score | -5.51 (0.43) | -5.09 (0.51)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Positive score: difference from placebo; Test type: Superiority or Other; p = 0.0412, ANCOVA — Mixed effects repeated measures (MMRM) analysis of covariance model with subject as random effect, treatment, region, visit, and visit-by-treatment interaction as fixed effects and baseline score as a covariate; Least squares mean = -1.33, 95% CI 2-sided [-2.61 to -0.05], Standard Error of Mean 0.65
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; Negative score: difference from placebo; Test type: Superiority or Other; p = 0.4661, ANCOVA — [p-value comment as in outcome 4, analysis 1]; Least squares mean = -0.43, 95% CI 2-sided [-1.57 to 0.72], Standard Error of Mean 0.58

5. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) Score at Week 6
Description: CGI-I: single-item clinician rated scale used to assess the subject's improvement or worsening from baseline. Scores range from 1 (very much improved) to 4 (no change) to 7 (very much worse); higher score indicates more affected.
Time Frame: Baseline, Week 6
Population: ITT; N=number of subjects with analyzable data at post-baseline observation.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 190 | 87
scores on a scale | 2.66 (0.09) | 2.85 (0.12)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Difference from placebo; Test type: Superiority or Other; p = 0.1820, ANOVA — Mixed effects MMRM with subject as random effect, treatment, region, visit and visit-by-treatment interaction as fixed effects; Least squares mean = -0.19, 95% CI 2-sided [-0.47 to 0.09], Standard Error of Mean 0.14

6. Secondary Outcome: Change From Baseline in Children's Global Assessment Scale (CGAS)
Description: CGAS: clinician-rated global assessment item for children based on symptoms and social functioning in home, school, and community settings. Scores on this single item range from 1 to 100 (higher levels indicate greater health) with descriptive anchors for every 10-point interval. Scores above 70 on this scale are considered within the "normal" range; lower score indicates need for increased supervision.
Time Frame: Baseline, Week 2, Week 4, Week 6, Early termination (ET)
Population: ITT; (n)=number of subjects with analyzable data at post-baseline observation for ziprasidone and placebo, respectively. ET includes observations from visits not within windowing criteria. Last observation carried forward [LOCF] imputation used for Week 6 LOCF timepoint.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 193 | 90
scores on a scale
  Week 2 (n=183, 86) | 4.7 (8.7) [3.4 to 5.9] | 2.6 (5.8) [1.3 to 3.8]
  Week 4 (n=155, 63) | 7.9 (10.4) [6.2 to 9.5] | 6.2 (8.9) [4.0 to 8.5]
  Week 6 (n=135, 52) | 10.9 (11.8) [8.9 to 12.9] | 10.8 (9.9) [8.0 to 13.5]
  ET (n=20, 15) | 1.3 (10.1) [-3.4 to 6.0] | 1.7 (8.9) [-3.2 to 6.6]
  Week 6 [LOCF] (n=185, 87) | 8.4 (11.8) [6.7 to 10.2] | 6.4 (10.6) [4.2 to 8.7]

7. Secondary Outcome: Change From Baseline in Child Health Questionnaire (CHQ)
Description: CHQ: 50-item, 15 subscale parent or legal guardian assessed instrument of child's physical, emotional, social well-being, and relative burden of disease on the parents; rated on Likert-type scale: range 0 to 100; higher scores indicate a more positive health status. Global indicators for Physical Health and Psychosocial Health are weighted composites derived from subscale items using scoring algorithms (transformed scores); range 0 to 100: higher scores indicate more positive health status.
Time Frame: Baseline, Week 6, ET
Population: ITT. ET includes observations from visits not within windowing criteria. LOCF imputation used for Week 6 LOCF timepoint.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 193 | 90
scores on a scale
  Global health: Week 6 | 5.0 (18.2) [2.0 to 8.1] | 8.5 (24.7) [1.5 to 15.5]
  Global health: ET | -5.4 (24.0) [-13.5 to 2.7] | -9.1 (17.4) [-15.3 to -2.8]
  Global health: Week 6 [LOCF] | 2.8 (19.9) [-0.1 to 5.8] | 1.4 (23.7) [-3.9 to 6.6]
  Global behavior: Week 6 | 9.4 (23.6) [5.4 to 13.4] | 10.9 (22.1) [4.6 to 17.2]
  Global behavior: ET | 6.4 (21.4) [-0.8 to 13.6] | -0.5 (23.0) [-8.8 to 7.8]
  Global behavior: Week 6 [LOCF] | 8.8 (23.1) [5.3 to 12.3] | 6.5 (23.1) [1.4 to 11.7]
  Family cohesion: Week 6 | 1.9 (21.3) [-1.7 to 5.6] | -0.8 (19.7) [-6.4 to 4.8]
  Family cohesion: ET | -1.8 (18.4) [-8.0 to 4.4] | -2.6 (16.1) [-8.5 to 3.3]
  Family cohesion: Week 6 [LOCF] | 1.2 (20.8) [-2.0 to 4.3] | -1.1 (18.1) [-5.2 to 2.9]
  Physical health: Week 6 | 3.5 (33.9) [-2.3 to 9.3] | 5.0 (28.0) [-3.0 to 13.0]
  Physical health: ET | -6.5 (32.9) [-17.6 to 4.7] | 3.2 (23.3) [-5.3 to 11.8]
  Physical health: Week 6 [LOCF] | 1.4 (33.8) [-3.8 to 6.5] | 4.8 (26.0) [-1.0 to 10.6]
  Bodily pain: Week 6 | 4.4 (21.6) [0.7 to 8.1] | 8.0 (19.4) [2.5 to 13.5]
  Bodily pain: ET | 4.7 (23.0) [-3.1 to 12.5] | 0.0 (14.6) [-5.3 to 5.3]
  Bodily pain: Week 6 [LOCF] | 4.5 (21.9) [1.2 to 7.8] | 4.9 (18.1) [0.9 to 8.9]
  Emotion, behavior: Week 6 | 16.2 (29.8) [11.0 to 21.3] | 13.8 (31.1) [4.9 to 22.6]
  Emotion, behavior: ET | 4.0 (43.1) [-10.6 to 18.6] | -2.5 (22.7) [-10.8 to 5.8]
  Emotion, behavior: Week 6 [LOCF] | 13.6 (33.4) [8.5 to 18.6] | 7.8 (29.2) [1.3 to 14.3]
  Time impact on parent: Week 6 | 8.8 (25.4) [4.5 to 13.1] | 11.8 (23.1) [5.2 to 18.4]
  Time impact on parent: ET | 2.0 (25.8) [-6.7 to 10.7] | 1.8 (21.7) [-6.2 to 9.7]
  Time impact on parent: Week 6 [LOCF] | 7.4 (25.5) [3.6 to 11.2] | 8.0 (23.1) [2.9 to 13.2]
  Emotional impact on parent: Week 6 | 8.9 (21.6) [5.2 to 12.5] | 10.0 (22.3) [3.7 to 16.3]
  Emotional impact on parent: ET | 3.5 (21.2) [-3.7 to 10.6] | 2.7 (12.6) [-1.8 to 7.3]
  Emotional impact on parent: Week 6 [LOCF] | 7.7 (21.6) [4.5 to 11.0] | 7.4 (19.4) [3.1 to 11.6]
  Mental health: Week 6 | 8.1 (15.3) [5.5 to 10.7] | 12.6 (18.2) [7.4 to 17.8]
  Mental health: ET | 1.3 (17.9) [-4.8 to 7.3] | -0.8 (12.0) [-5.2 to 3.6]
  Mental health: Week 6 [LOCF] | 6.7 (16.1) [4.2 to 9.1] | 7.5 (17.4) [3.6 to 11.4]
  Physical function: Week 6 | 5.6 (19.7) [2.2 to 8.9] | 5.9 (25.2) [-1.3 to 13.1]
  Physical function: ET | -5.4 (22.5) [-13.0 to 2.2] | -0.2 (17.7) [-6.6 to 6.2]
  Physical function: Week 6 [LOCF] | 3.3 (20.8) [0.2 to 6.4] | 3.7 (22.8) [-1.3 to 8.7]
  Behavior scale: Week 6 | 9.0 (17.1) [6.1 to 11.9] | 9.0 (16.8) [4.2 to 13.8]
  Behavior scale: ET | 7.6 (15.2) [2.4 to 12.9] | 0.6 (17.1) [-5.6 to 6.7]
  Behavior scale: Week 6 [LOCF] | 8.7 (16.7) [6.2 to 11.3] | 5.8 (17.4) [1.9 to 9.6]
  Self-esteem: Week 6 | 6.0 (17.5) [3.1 to 9.0] | 9.0 (22.9) [2.5 to 15.5]
  Self-esteem: ET | 1.0 (20.6) [-5.9 to 8.0] | 1.3 (14.0) [-3.8 to 6.5]
  Self-esteem: Week 6 [LOCF] | 5.0 (18.2) [2.3 to 7.7] | 6.4 (20.2) [1.9 to 10.9]
  General health perception: Week 6 | 1.1 (11.6) [-0.9 to 3.1] | 3.3 (11.7) [0.0 to 6.7]
  General health perception: ET | -2.2 (12.3) [-6.3 to 2.0] | -0.6 (10.8) [-4.5 to 3.3]
  General health perception: Week 6 [LOCF] | 0.4 (11.8) [-1.3 to 2.2] | 1.8 (11.5) [-0.8 to 4.3]
  Family activities: Week 6 | 9.2 (22.6) [5.3 to 13.0] | 14.6 (22.5) [8.2 to 21.0]
  Family activities: ET | 1.3 (16.8) [-4.5 to 7.1] | -4.6 (16.5) [-10.6 to 1.5]
  Family activities: Week 6 [LOCF] | 7.5 (21.7) [4.3 to 10.8] | 7.8 (22.0) [2.9 to 12.7]
  Change in health: Week 6 | 0.5 (1.1) [0.3 to 0.6] | 0.6 (1.0) [0.3 to 0.9]
  Change in health: ET | -0.4 (1.0) [-0.7 to -0.1] | -0.1 (0.8) [-0.4 to 0.2]
  Change in health: Week 6 [LOCF] | 0.3 (1.1) [0.1 to 0.5] | 0.3 (1.0) [0.1 to 0.6]
  Physical health global subscale: Week 6 | 1.8 (9.7) [0.2 to 3.5] | 2.4 (9.8) [-0.4 to 5.2]
  Physical health global subscale: ET | -2.8 (11.8) [-6.9 to 1.3] | 0.1 (4.4) [-1.5 to 1.7]
  Physical health global subscale: Week 6 [LOCF] | 0.9 (10.3) [-0.7 to 2.4] | 1.6 (8.2) [-0.2 to 3.4]
  Psychosocial health global subscale: Week 6 | 6.6 (9.5) [5.0 to 8.3] | 7.7 (11.0) [4.5 to 10.9]
  Psychosocial health global subscale: ET | 3.1 (10.4) [-0.5 to 6.6] | 0.0 (5.7) [-2.0 to 2.1]
  Psychosocial health global subscale: Week 6 [LOCF] | 5.9 (9.8) [4.4 to 7.4] | 4.8 (10.0) [2.6 to 7.1]

8. Secondary Outcome: Change From Baseline in Children's Problem Behavior and Aggression Questionnaire (CPBAQ) Total Score
Description: CPBAQ: 19-item parent or legal guardian completed questionnaire to rate the child's verbal (such as yelling or cursing) and physical aggression (such a fighting with peers or being cruel to an animal) during the past week. Behavior was rated on a 4-point scale; range 0 (behavior did not occur or was not a problem) to 3 (behavior occurred a lot or was severe problem). Total score range 0 to 57; higher scores indicate a greater frequency and severity of aggression.
Time Frame: Baseline, Week 1 through Week 6
Population: ITT; N=number of subjects with analyzable data at baseline; (n)= number of subjects with analyzable data at post-baseline observation for ziprasidone and placebo, respectively. LOCF imputation used for Week 6 LOCF timepoint.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 173 | 74
scores on a scale
  Week 1 (n=165, 69) | -2.4 (7.1) [-3.53 to -1.33] | -1.3 (5.8) [-2.72 to 0.05]
  Week 2 (n=161, 71) | -2.5 (8.0) [-3.79 to -1.29] | -1.0 (6.2) [-2.42 to 0.51]
  Week 3 (n=146, 64) | -3.0 (6.7) [-4.06 to -1.88] | -0.7 (5.7) [-2.08 to 0.77]
  Week 4 (n=138, 51) | -2.7 (7.4) [-3.96 to -1.46] | -1.0 (6.5) [-2.79 to 0.87]
  Week 5 (n=126, 44) | -3.1 (7.0) [-4.32 to -1.86] | -0.8 (8.3) [-3.32 to 1.73]
  Week 6 (n=119, 42) | -3.0 (7.4) [-4.30 to -1.62] | -1.9 (6.7) [-3.94 to 0.22]
  Week 6 [LOCF] (n=167, 71) | -2.3 (8.2) [-3.58 to -1.07] | -0.3 (8.8) [-2.37 to 1.81]

9. Secondary Outcome: Change From Baseline in Child Depression Rating Scale - Revised (CDRS-R): Total Score
Description: CDRS-R: clinician-rated interview-based scale (with both child and parent or guardian) to assess 17 distinct symptom areas to derive an index of depression severity. Discrepancies between informants' responses were resolved by using most impaired rating given by valid informant. Rated on a 7-point scale; range from 1 (no impairment) to 7 (indicates greater impairment). Total score calculated as sum of the 17 items (range 1 to 119); higher score indicates greater impairment.
Time Frame: Baseline, Week 1 through Week 6
Population: ITT; N=number of subjects with analyzable data at baseline; (n)=number of subjects with analyzable data at post-baseline observation for ziprasidone and placebo, respectively. LOCF imputation used for Week 6 LOCF timepoint.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 180 | 84
scores on a scale
  Week 1 (n=179, 82) | -2.8 (6.6) [-3.78 to -1.84] | -1.4 (5.7) [-2.62 to -0.11]
  Week 2 (n=174, 80) | -4.2 (7.3) [-5.24 to -3.07] | -2.5 (5.6) [-3.73 to -1.25]
  Week 3 (n=157, 69) | -5.5 (7.4) [-6.69 to -4.35] | -3.2 (5.4) [-4.48 to -1.90]
  Week 4 (n=148, 59) | -6.0 (7.6) [-7.20 to -4.74] | -4.9 (6.6) [-6.65 to -3.18]
  Week 5 (n=135, 49) | -7.0 (8.5) [-8.47 to -5.57] | -5.6 (5.9) [-7.30 to -3.92]
  Week 6 (n=126, 47) | -7.9 (7.9) [-9.29 to -6.52] | -6.5 (5.5) [-8.13 to -4.89]
  Week 6 [LOCF] (n=178, 82) | -5.8 (8.7) [-7.07 to -4.51] | -4.0 (7.3) [-5.64 to -2.43]

10. Secondary Outcome: Change From Baseline in Child Depression Rating Scale - Revised (CDRS-R): Suicide Ideation Item 13
Description: CDRS-R: clinician-rated interview-based scale (with both child and parent or guardian) to assess 17 distinct symptom areas to derive an index of depression severity. Discrepancies between informants' responses were resolved by using most impaired rating given by valid informant. Suicide Ideation (Item 13) detects changes in suicidality over time. Rated on a 7-point scale; range from 1 (no impairment) to 7 (indicates greater impairment).
Time Frame: Baseline, Week 1 through Week 6
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 192 | 90
scores on a scale
  Week 1 (n=188, 86) | -0.1 (0.4) | -0.0 (0.5)
  Week 2 (n=182, 86) | -0.0 (0.5) | -0.1 (0.5)
  Week 3 (n=165, 74) | -0.1 (0.5) | -0.1 (0.3)
  Week 4 (n=154, 63) | 0.0 (0.5) | -0.1 (0.5)
  Week 5 (n=141, 54) | 0.0 (0.4) | -0.1 (0.5)
  Week 6 (n=134, 52) | -0.0 (0.3) | -0.1 (0.4)
  Week 6 [LOCF] (n=189, 87) | 0.0 (0.6) | -0.0 (0.5)

11. Secondary Outcome: Change From Baseline in Child Depression Rating Scale - Revised (CDRS-R): Impaired Schoolwork Item 1
Description: Clinician-rated interview-based scale (with both child and parent or guardian) to assess 17 distinct symptom areas to derive an index of depression severity. Discrepancies between informants' responses resolved by using most impaired rating given by valid informant. Impaired Schoolwork (Item 1) assesses school function for the subgroup of subjects reported to be in school. Rated on a 7-point scale; range from 1 (no impairment) to 7 (indicates greater impairment).
Time Frame: Baseline, Week 2, Week 6
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 40 | 15
scores on a scale
  Week 2 (n=38, 15) | -0.3 (0.9) | -0.2 (0.7)
  Week 6 (n=30, 8) | -0.6 (1.1) | -0.1 (1.4)
  Week 6 [LOCF] (n=39, 15) | -0.6 (1.0) | -0.1 (1.1)

12. Secondary Outcome: Change From Baseline in CNS Vital Signs Cognitive Test Battery (Includes Sedation Item): Subscales
Description: A computerized subject-administered test battery with subtests for verbal and visual memory, processing speed, nonverbal reasoning, executive functioning, working memory, and sustained attention. A computerized 7-point sedation item (0 [not sleepy] to 10 [very sleepy]) was completed prior to test battery. The Neurocognitive index score was derived from subtest scores per an algorithm. The index score and subtest scores assessed the subject's changes in cognition. Scores were rated as above average (score >109), average (90 to 109), below average (80 to 89), or well below average (70 to 79).
Time Frame: Baseline, Week 6, ET
Population: ITT; N=number of subjects with analyzable data at baseline; (n)= number of subjects with analyzable data at post-baseline observation for ziprasidone and placebo, respectively. ET includes observations from visits not within windowing criteria. LOCF imputation used for Week 6 LOCF timepoint (last post-baseline non-missing visit).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 174 | 83
scores on a scale
  Sedation: Week 6 (n=124, 47) | 0.0 (1.7) [-0.27 to 0.33] | -0.4 (1.8) [-0.98 to 0.08]
  Sedation: ET (n=23, 26) | 0.0 (2.3) [-0.98 to 0.98] | 0.2 (1.3) [-0.34 to 0.73]
  Sedation: Week 6 [LOCF] (n=147, 72) | 0.0 (1.8) [-0.28 to 0.30] | -0.2 (1.7) [-0.63 to 0.16]
  Verbal Memory: Week 6 (n=124, 47) | 1.3 (12.1) [-0.83 to 3.45] | 0.5 (14.0) [-3.63 to 4.59]
  Verbal Memory: ET (n=24, 25) | -2.3 (13.9) [-8.22 to 3.53] | -2.6 (15.1) [-8.80 to 3.66]
  Verbal Memory: Week 6 [LOCF] (n=148, 71) | 0.7 (12.4) [-1.39 to 2.66] | -0.5 (14.4) [-3.95 to 2.87]
  Visual Memory: Week 6 (n=124, 46) | 0.5 (13.3) [-1.89 to 2.83] | 2.0 (14.5) [-2.31 to 6.28]
  Visual Memory: ET (n=24, 26) | -3.8 (10.2) [-8.10 to 0.48] | 0.4 (14.2) [-5.28 to 6.17]
  Visual Memory: Week 6 [LOCF] (n=148, 71) | -0.2 (12.9) [-2.46 to 1.69] | 1.2 (14.3) [-2.19 to 4.60]
  Processing Speed: Week 6 (n=124, 46) | 1.3 (13.5) [-1.06 to 3.73] | 1.0 (12.0) [-2.58 to 4.53]
  Processing Speed: ET (n=24, 25) | -10.6 (34.5) [-25.14 to 3.99] | 0.5 (5.4) [-1.73 to 2.74]
  Processing Speed: Week 6 [LOCF] (n=148, 70) | -0.6 (18.9) [-3.73 to 2.45] | 0.6 (10.1) [-1.76 to 3.06]
  Reasoning: Week 6 (n=122, 46) | 2.2 (12.0) [0.09 to 4.41] | -0.7 (14.6) [-5.03 to 3.65]
  Reasoning: ET (n=23, 25) | 1.3 (15.8) [-5.56 to 8.12] | 3.3 (14.0) [-2.47 to 9.13]
  Reasoning: Week 6 [LOCF] (n=145, 70) | 1.9 (12.7) [-0.16 to 4.03] | 0.7 (14.1) [-2.66 to 4.06]
  Executive Functioning: Week 6 (n=123, 46) | 2.9 (15.4) [0.19 to 5.68] | 2.7 (18.2) [-2.76 to 8.07]
  Executive Functioning: ET (n=23, 26) | -6.7 (9.1) [-10.61 to -2.77] | 4.6 (13.2) [-0.68 to 9.95]
  Executive Functioning: Week 6 [LOCF] (n=146, 71) | 1.4 (14.9) [-1.04 to 3.88] | 3.2 (16.6) [-0.71 to 7.14]
  Working Memory: Week 6 (n=120, 45) | 1.9 (12.9) [-0.40 to 4.26] | 0.5 (12.9) [-3.32 to 4.41]
  Working Memory: ET (n=23, 24) | 3.2 (13.5) [-2.66 to 9.03] | 3.7 (11.0) [-0.93 to 8.39]
  Working Memory: Week 6 [LOCF] (n=143, 68) | 2.0 (12.9) [-0.20 to 4.10] | 1.3 (12.2) [-1.64 to 4.27]
  Sustained Attention: Week 6 (n=120, 45) | 2.0 (12.3) [-0.18 to 4.26] | -1.6 (13.1) [-5.59 to 2.30]
  Sustained Attention: ET (n=23, 24) | 0.5 (13.5) [-5.27 to 6.37] | 1.5 (11.6) [-3.42 to 6.37]
  Sustained Attention: Week 6 [LOCF] (n=143, 68) | 1.7 (12.4) [-0.54 to 3.47] | -0.9 (12.6) [-3.98 to 2.10]

13. Secondary Outcome: Change From Baseline in CNS Vital Signs Cognitive Test Battery: Neurocognitive Index
Description: as for outcome 12
Time Frame: Baseline, Week 6, ET
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 168 | 79
scores on a scale
  Neurocognitive Index: Week 6 (n=120, 45) | 1.8 (7.1) | 0.8 (7.5)
  Neurocognitive Index: ET (n=23, 23) | -2.7 (7.6) | 2.2 (7.2)
  Neurocognitive Index: Week 6 [LOCF] (n=143, 67) | 1.0 (7.4) | 1.1 (7.4)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Neurocognitive Index score at Week 6: difference from placebo; Test type: Superiority or Other; p = 0.2613, ANCOVA — SAS PROC MIXED to fit a mixed model analysis of covariance with treatment and region as fixed effects and baseline score as covariate; Observed cases at Week 6; Least squares mean = 1.34, 95% CI 2-sided [-1.01 to 3.69], Standard Error of Mean 1.19

14. Secondary Outcome: Change From Baseline in Movement Disorder Scales: Simpson-Angus Rating Scale (SARS)
Description: SARS: 10-item clinician rated instrument to assess parkinsonian symptoms (7 items) and related extrapyramidal side effects (3 items): gait, arm dropping, shoulder shaking, elbow rigidity, leg pendulousness, glabellar tap, tremor, and salivation. Head dropping (modified SARS item 7) substituted for head rotation. Anchored 5-point scale: range 0 (absence of condition, normal) to 4 (most extreme form of condition). Total score is sum of individual item scores (range 0 to 40); higher score indicates more affected.
Time Frame: Baseline, Week 1 through Week 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 189 | 87
scores on a scale
  Week 1 (n=189, 85) | 0.5 (2.8) [0.12 to 0.93] | 0.1 (0.9) [-0.10 to 0.29]
  Week 2 (n=182, 85) | 0.5 (2.4) [0.17 to 0.88] | -0.0 (0.5) [-0.13 to 0.08]
  Week 3 (n=165, 74) | 0.7 (3.1) [0.18 to 1.15] | 0.3 (1.6) [-0.09 to 0.65]
  Week 4 (n=154, 62) | 0.4 (2.6) [-0.01 to 0.83] | -0.0 (0.6) [-0.20 to 0.11]
  Week 5 (n=141, 54) | 0.2 (2.4) [-0.18 to 0.63] | -0.0 (1.0) [-0.30 to 0.26]
  Week 6 (n=134, 52) | 0.2 (2.5) [-0.27 to 0.58] | -0.2 (0.8) [-0.37 to 0.06]
  Week 6 [LOCF] (n=189, 86) | 0.3 (2.5) [-0.09 to 0.63] | -0.1 (0.6) [-0.21 to 0.07]

15. Secondary Outcome: Change From Baseline in Movement Disorder Scales: Barnes Akathisia Rating Scale (BAS) Global Clinical Assessment Item
Description: BAS: clinician rated scale to assess akathisia to determine the degree of subjective restlessness and distress associated with restlessness. First 3 items (Objective, Subjective, and Distress related to restlessness) rated on a 4-point scale with range 0 (no symptoms) to 3 (increased severity of symptoms). Item 4 Global Clinical Assessment of Akathisia rated on a 6-point scale range 0 (no symptoms) to 5 (increased severity of symptoms); higher score indicates increased severity. All rating are anchored. Only the Global Clinical Assessment of Akathisia was to be analyzed.
Time Frame: Baseline, Week 1 through Week 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 190 | 88
scores on a scale
  Week 1 (n=190, 86) | 0.1 (0.6) [-0.03 to 0.15] | 0.1 (0.4) [0.01 to 0.20]
  Week 2 (n=183, 86) | 0.1 (0.7) [0.02 to 0.22] | 0.0 (0.3) [-0.05 to 0.07]
  Week 3 (n=166, 74) | 0.1 (0.6) [-0.04 to 0.15] | 0.0 (0.3) [-0.02 to 0.10]
  Week 4 (n=155, 63) | 0.1 (0.6) [-0.03 to 0.15] | -0.0 (0.2) [-0.08 to 0.01]
  Week 5 (n=142, 54) | 0.1 (0.5) [-0.03 to 0.15] | 0.0 (0.2) [-0.05 to 0.05]
  Week 6 (n=135, 52) | 0.0 (0.5) [-0.06 to 0.11] | 0.0 (0.2) [-0.06 to 0.06]
  Week 6 [LOCF] (n=190, 87) | 0.0 (0.6) [-0.08 to 0.08] | 0.0 (0.2) [-0.04 to 0.06]

16. Secondary Outcome: Change From Baseline in Movement Disorder Scales: Abnormal Involuntary Movement Scale (AIMS) Movement Cluster Score
Description: AIMS: clinician rated 12-item scale to rate 7 body areas and global judgments on the severity of abnormal movements, incapacitation and subject's awareness of abnormal movements. Items 1 to 10 scored 0 (none) to 4 (severe) (total possible score 0 to 40; higher score indicates greater severity); items 11 to 14 are No or Yes response to dental status and sleep movements. Only the sum of the first 7 items to be analyzed (AIMS Movement Cluster score). Total score 0 to 28; higher score indicates greater severity.
Time Frame: Baseline, Week 1 through Week 6
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 190 | 88
scores on a scale
  Week 1 (n=190, 86) | 0.2 (1.6) [-0.04 to 0.42] | -0.0 (0.4) [-0.10 to 0.06]
  Week 2 (n=183, 86) | 0.1 (1.6) [-0.09 to 0.37] | 0.0 (0.6) [-0.10 to 0.17]
  Week 3 (n=166, 74) | 0.1 (1.3) [-0.12 to 0.28] | 0.1 (1.0) [-0.08 to 0.37]
  Week 4 (n=155, 63) | 0.1 (0.8) [-0.07 to 0.18] | -0.0 (0.8) [-0.23 to 0.17]
  Week 5 (n=142, 54) | -0.1 (0.7) [-0.18 to 0.05] | 0.0 (0.4) [-0.12 to 0.12]
  Week 6 (n=135, 52) | 0.0 (0.6) [-0.11 to 0.11] | 0.0 (0.5) [-0.15 to 0.15]
  Week 6 [LOCF] (n=190, 87) | 0.0 (0.8) [-0.11 to 0.11] | -0.0 (0.7) [-0.18 to 0.14]

17. Secondary Outcome: Number of Subjects Per Response on the School Placement Questionnaire: School Situation
Description: School placement questionnaire: parent or legal guardian assessed questionnaire to determine whether the child is currently enrolled in school (or planned to be enrolled if on school holiday like summer break), whether attending regularly if enrolled, and how well the child is doing overall in school. Questions were modified from those used in the National Institute of Mental Health (NIMH) funded Treatment of Early Onset Schizophrenia Spectrum (TEOSS) study. Results determine whether subjects are currently attending school and qualitatively describe how well they are doing in school.
Time Frame: Baseline, Week 2, Week 6, ET
Population: ITT; N=number of subjects analyzable for School Placement Questionnaire; (n)=number of subjects with analyzable data at baseline and post-baseline observation for ziprasidone and placebo, respectively. ET includes observations from visits not within windowing criteria. LOCF imputation used for Week 6 LOCF timepoint.
Measure: Number; unit: participants
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 189 | 87
participants
  Baseline: Enrolled or attend (n=185, 85) | 40 | 15
  Baseline: Not attend or mental illness (n=185, 85) | 62 | 26
  Baseline: Not attend or other (n=185, 85) | 2 | 0
  Baseline: Enrolled or vacation (n=185, 85) | 20 | 19
  Baseline: Not enrolled or mental illness | 36 | 12
  Baseline: Not enrolled or other (n=185, 85) | 25 | 13
  Week 2: Enrolled or attend (n=179, 84) | 38 | 20
  Week 2: Not attend or mental illness (n=179, 84) | 59 | 24
  Week 2: Not attend or other (n=179, 84) | 3 | 2
  Week 2: Enrolled or vacation (n=179, 84) | 20 | 11
  Week 2: Not enrolled or mental illness (n=179, 84) | 36 | 15
  Week 2: Not enrolled or other (n=179, 84) | 23 | 12
  Week 6: Enrolled or attend (n=134, 51) | 38 | 18
  Week 6: Not attend or mental illness (n=134, 51) | 36 | 7
  Week 6: Not attend or other (n=134, 51) | 3 | 0
  Week 6: Enrolled or vacation (n=134, 51) | 14 | 5
  Week 6: Not enrolled or mental illness (n=134, 51) | 23 | 11
  Week 6: Not enrolled or other (n=134, 51) | 20 | 10
  ET: Enrolled or attend (n=32, 25) | 5 | 3
  ET: Not attend or mental illness (n=32, 25) | 8 | 14
  ET: Not attend or other (n=32, 25) | 0 | 0
  ET: Enrolled or vacation (n=32, 25) | 5 | 4
  ET: Not enrolled or mental illness (n=32, 25) | 10 | 3
  ET: Not enrolled or other (n=32, 25) | 4 | 1
  Week 6 [LOCF]: Enrolled or attend (n=183, 86) | 47 | 23
  Week 6 [LOCF]: Not attend or mental illness | 50 | 86
  Week 6 [LOCF]: Not attend or other (n=183, 86) | 3 | 1
  Week 6 [LOCF]: Enrolled or vacation (n=183, 86) | 21 | 10
  Week 6 [LOCF]: Not enrolled or mental illness | 36 | 17
  Week 6 [LOCF]: Not enrolled or other (n=183, 86) | 26 | 12

18. Secondary Outcome: Number of Subjects Per Response on the School Placement Questionnaire: School Attendance
Description: as for outcome 17
Time Frame: Baseline, Week 2, Week 6, ET
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 189 | 87
participants
  Baseline: No absences (n=88, 42) | 20 | 7
  Baseline: Only a few absences (n=88, 42) | 16 | 15
  Baseline: Frequent absences (n=88, 42) | 13 | 2
  Baseline: Did not attend (n=88, 42) | 26 | 7
  Baseline: Not applicable or vacation (n=88, 42) | 13 | 11
  Week 2: No absences (n=82, 36) | 19 | 8
  Week 2: Only a few absences (n=82, 36) | 14 | 9
  Week 2: Frequent absences (n=82, 36) | 11 | 4
  Week 2: Did not attend (n=82, 36) | 25 | 8
  Week 2: Not applicable or vacation (n=82, 36) | 13 | 7
  Week 6: No absences (n=67, 24) | 16 | 8
  Week 6: Only a few absences (n=67, 24) | 22 | 12
  Week 6: Frequent absences (n=67, 24) | 5 | 0
  Week 6: Did not attend (n=67, 24) | 13 | 0
  Week 6: Not applicable or vacation (n=67, 24) | 11 | 4
  ET: No absences (n=12, 12) | 1 | 0
  ET: Only a few absences (n=12, 12) | 4 | 0
  ET: Frequent absences (n=12, 12) | 2 | 5
  ET: Did not attend (n=12, 12) | 4 | 4
  ET: Not applicable or vacation (n=12, 12) | 1 | 3
  Week 6 [LOCF]: No absences (n=89, 37) | 18 | 8
  Week 6 [LOCF]: Only a few absences (n=89, 37) | 26 | 13
  Week 6 [LOCF]: Frequent absences (n=89, 37) | 11 | 4
  Week 6 [LOCF]: Did not attend (n=89, 37) | 21 | 4
  Week 6[LOCF]: Not applicable or vacation(n=89,37) | 13 | 8

19. Secondary Outcome: Number of Subjects Per Response on the School Placement Questionnaire: Overall School Performance
Description: as for outcome 17
Time Frame: Baseline, Week 2, Week 6, ET
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 189 | 87
participants
  Baseline: Excellent (n=64, 29) | 4 | 2
  Baseline: Good (n=64, 29) | 10 | 6
  Baseline: Fair (n=64, 29) | 25 | 14
  Baseline: Poor (n=64, 29) | 19 | 3
  Baseline: Very poor (n=64, 29) | 6 | 4
  Week 2: Excellent (n=60, 26) | 5 | 1
  Week 2: Good (n=60, 26) | 12 | 8
  Week 2: Fair (n=60, 26) | 20 | 10
  Week 2: Poor (n=60, 26) | 17 | 5
  Week 2: Very poor (n=60, 26) | 6 | 2
  Week 6: Excellent (n=52, 21) | 4 | 1
  Week 6: Good (n=52, 21) | 16 | 8
  Week 6: Fair (n=52, 21) | 17 | 11
  Week 6: Poor (n=52, 21) | 12 | 1
  Week 6: Very poor (n=52, 21) | 3 | 0
  ET: Excellent (n=8, 7) | 0 | 0
  ET: Good (n=8, 7) | 0 | 1
  ET: Fair (n=8, 7) | 5 | 3
  ET: Poor (n=8, 7) | 2 | 1
  ET: Very poor (n=8, 7) | 1 | 2
  Week 6 [LOCF]: Excellent (n=68, 28) | 4 | 1
  Week 6 [LOCF]: Good (n=68, 28) | 18 | 9
  Week 6 [LOCF]: Fair (n=68, 28) | 24 | 14
  Week 6 [LOCF]: Poor (n=68, 28) | 16 | 2
  Week 6 [LOCF]: Very poor (n=68, 28) | 6 | 2

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events are reported from time of first dose of study treatment up to 6 days after last dose of study treatment.
Description: Safety population = all randomized subjects with at least 1 dose of study treatment. An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and = non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event.
Arm/Group | Ziprasidone | Placebo
Serious Adverse Events (participants affected / at risk) | 9/193 | 1/90
Other Adverse Events (participants affected / at risk) | 110/193 | 27/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=193) | Placebo (N=90)
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Aggression (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 1 | 0
Hostility (Psychiatric disorders) | 1 | 0
Impulsive behaviour (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 2 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=193) | Placebo (N=90)
Nausea (Gastrointestinal disorders) | 19 | 2
Vomiting (Gastrointestinal disorders) | 12 | 3
Fatigue (General disorders) | 17 | 4
Overdose (Injury, poisoning and procedural complications) | 11 | 4 — All overdoses were due to clinical or subject error.
Akathisia (Nervous system disorders) | 13 | 3
Dizziness (Nervous system disorders) | 18 | 1
Extrapyramidal disorder (Nervous system disorders) | 22 | 1
Headache (Nervous system disorders) | 15 | 2
Somnolence (Nervous system disorders) | 38 | 6
Tremor (Nervous system disorders) | 15 | 1
Insomnia (Psychiatric disorders) | 18 | 13

LIMITATIONS AND CAVEATS:
The AE tables were amended to incorporate previously unreported AEs that were found during an independent audit and verified by the investigators.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.